CLINICAL TRIAL: NCT03655808
Title: Autologous Transplantation of Bronchial Basal Cells for Treatment of Bronchiectasis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Collaborators: Regend Therapeutics (Industry)
Responsible Party: Principal Investigator, Jieming QU, Principal Investigator, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201810
Record Dates: First submitted 2018-08-22; First posted 2018-08-31 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Bronchiectasis
Keywords: Bronchiectasis; Bronchial basal cells; Autologous transplantation
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Intervention Model Description: Eligibility patients were randomly assigned in a 1:1 ratio to receive either autologous cell transplantation therapy (cell treatment group) or bronchoscopic airway clearance treatment (B-ACT therapy, control group).
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The opaque sealed envelope method was used to conceal the allocation sequence. Both patients and investigators, except for the bronchoscopy operators, remained masked to the treatment assignment for the duration of the study. Only the investigators who performed the bronchoscopy were unblinded. The non-blinded investigators should not disclose any blind information to other investigators, participants, care providers, or outcomes assessors.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cell treatment group (Experimental): Patients receive both autologous BBCs transplantation and B-ACT therapy.
  Interventions: Biological: Bronchial basal cells (BBCs); Procedure: Bronchoscopic airway clearance treatment （B-ACT）
- Control group (Sham Comparator): Patients only receive B-ACT therapy.
  Interventions: Procedure: Bronchoscopic airway clearance treatment （B-ACT）

INTERVENTIONS:
Biological: Bronchial basal cells (BBCs) — Airway epithelial cells were collected in patients of the cell treatment group by a disposable 2-mm brush in order to obtain BBCs. The obtained tissue were washed and enzymatically digested to form a single-cell suspension, which was then cultured under R-Clone system, a patented technique of Regend Therapeutics, Ltd.. For patients in the cell treatment group, on the basis of B-ACT therapy, they were also received autologous BBCs transplantation. Cell suspension was diluted with normal saline. Fibrotic bronchoscopy was guided into the lobular or segmental airways and cells were instilled into lobes.
  Other Names: P63+ lung stem/progenitor cells; Airway basal cells; Lung stem/progenitor cells
  Arms: Cell treatment group
Procedure: Bronchoscopic airway clearance treatment （B-ACT） — The bronchoscopy was performed by board-certified respiratory physicians of Ruijin Hospital using a flexible fiber-optic bronchoscope. B-ACT therapy was performed on all patients in both groups according to the protocol. In brief, continuous suction was performed with the sputum aspirator from the trachea to the subsegmental during the entering of bronchoscope to remove the visible secretions from entire respiratory tract, and then operators used normal saline to collect lavage fluid (the volume various depending on the operator's judgement).

SUMMARY:
Bronchiectasis is a disease resulted from progressive destruction of bronchi with no effective drug for its treatment. In this study, we intends to carry out a randomized, single-blinded, controlled pilot clinical trial at 1/2 phase. During the process, autologous bronchial basal cells (BBCs) will be dissected from trial tissue via bronchoscopic brushing. Then the BBCs will be expanded and detected by quality control. In the following, qualified BBCs will be injected directly into the lesion by fiberoptic bronchoscopy after airway clearance. The investigators will evaluate the safety and effectiveness of the treatment by measuring a serial of indicators, including occurrence of adverse events, pulmonary function, 6 minute walk distance (6MWD), the distance-saturation product (DSP), St. George's Respiratory Questionnaire (SGRQ), FACED scoring, bronchiectasis severity index (BSI) , and high-resolution computed tomography (HRCT) at week 4, week 12, and week 24 after cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed as bronchiectasis.
* Subjects with a DLCO < 80% predicted value.
* Subjects with stable condition for more than 2 weeks.
* Subjects can do pulmonary function tests.
* Subjects can tolerate bronchoscopy.
* Subjects signed informed consent.

Exclusion Criteria:

* Women of childbearing age at the stage of pregnancy or lactation, or those without taking effective contraceptive measures.
* Subjects with positive serological tests for hepatitis B virus (HBV), hepatitis C virus (HCV), human immunodeficiency virus (HIV) or syphilis (HBV carriers and patients with stable chronic hepatitis B could be accepted if titers of HBV DNA < 500 IU/mL or copies < 1000 copies/mL; patients with curative hepatitis C were eligible if HCV RNA tests were negative).
* Subjects with any malignancy.
* Subjects with any of the following pulmonary diseases: active tuberculosis, pulmonary embolism, pneumothorax, multiple huge bullae, uncontrolled asthma, acute exacerbation of chronic bronchitis or extremely severe COPD.
* Subjects with other serious diseases, such as poorly controlled diabetes, myocardial infarction, unstable angina, cirrhosis, and acute glomerulonephritis.
* Subjects with leukopenia (WBC less than 4x10^9 / L) or agranulocytosis (WBC less than 1.5x10^9 / L or neutrophils less than 0.5x10^9 / L) caused by any reason.
* Subjects with severe renal impairment, serum creatinine> 1.5 times of the upper limit of normal.
* Subjects with liver disease or liver damage: ALT, AST, total bilirubin> 2 times of the upper limit of normal.
* Subjects with a history of mental illness or suicide risk, with a history of epilepsy or other central nervous system disorders.
* Subjects with severe arrhythmias (such as ventricular tachycardia, frequent superventricular tachycardia, atrial fibrillation, and atrial flutter, etc.) or cardiac degree II or above conduction abnormalities displayed via 12-lead ECG.
* Subjects with a history of alcohol or illicit drug abuse.
* Subjects accepted by any other clinical trials within 3 months before the enrollment.
* Subjects with poor compliance, difficult to complete the study.
* Any other conditions that might increase the risk of subjects or interfere with the clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2020-06-21 (Actual); Primary Completion 2023-05-17 (Actual); Study Completion 2023-05-17 (Actual)

PRIMARY OUTCOMES:
Diffusing capacity of the lung for carbon monoxide (DLCO) | Week 4, 12, and 24 after treatment
  An indicator of pulmonary function

SECONDARY OUTCOMES:
Forced expiratory volume measured at the first second (FEV1) | Week 4, 12, and 24 after treatment
  An indicator for pulmonary function test to assess airway obstruction
Forced vital capacity (FVC) | Week 4, 12, and 24 after treatment
  An indicator for pulmonary function test to indicate the maximum amount of air a person can expel from the lungs after a maximum inhalation
The ratio of forced expiratory volume in the first one second to the forced vital capacity (FEV1/FVC) | Week 4, 12, and 24 after treatment
  An indicator in pulmonary function test to represent the proportion of a person's vital capacity that they are able to expire in the first second of forced expiration to the full vital capacity
Maximum Mid Expiratory Flow (MMEF) | Week 4, 12, and 24 after treatment
  An indicator in pulmonary function test to stand for maximal (mid-)expiratory flow and is the peak of expiratory flow as taken from the flow-volume curve and measured in liters per second
Maximum Voluntary Ventilation (MVV) | Week 4, 12, and 24 after treatment
  An indicator in pulmonary function test to measure the maximum amount of air that can be inhaled and exhaled within one minute
6 minute walk distance (6MWD) and distance saturation product (DSP) | Week 4, 12, and 24 after treatment
  An indicator for heart and pulmonary function
St. George's Respiratory Questionnaire (SGRQ) | Week 4, 12, and 24 after treatment
  An indicator to measure health status (quality of life) in patients with diseases of airways obstruction
FACED scoring | Week 4, 12, and 24 after treatment
  An assessment of severity tool, validated for people with non-cystic fibrosis bronchiectasis. F means "FEV1", A means "Age", C means "Chronic colonization", E means "Extension", D means "Dyspnoea".
Bronchiectasis Severity Index (BSI) | Week 4, 12, and 24 after treatment
  A combination of clinical, radiological and microbiological features to predict morbidity and mortality.
High resolution computed tomography (HR-CT) imaging of lung | Week 4, 12, and 24 after treatment
  An indicator for analysis of dilated bronchi, HR-CT images of lung will be analyzed to indicate the pulmonary structure
Safety outcomes: adverse events | Through study completion, an average of 24 weeks
  Any unexpected and unfavorable medical occurrence related to any medical intervention in the study

CONTACTS AND LOCATIONS:
Overall Officials: Yun Feng, M.D., Ph.D, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital Shanghai JiaoTong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zuo W, Zhang T, Wu DZ, Guan SP, Liew AA, Yamamoto Y, Wang X, Lim SJ, Vincent M, Lessard M, Crum CP, Xian W, McKeon F. p63(+)Krt5(+) distal airway stem cells are essential for lung regeneration. Nature. 2015 Jan 29;517(7536):616-20. doi: 10.1038/nature13903. Epub 2014 Nov 12. PMID 25383540
- [Background] Ma Q, Ma Y, Dai X, Ren T, Fu Y, Liu W, Han Y, Wu Y, Cheng Y, Zhang T, Zuo W. Regeneration of functional alveoli by adult human SOX9+ airway basal cell transplantation. Protein Cell. 2018 Mar;9(3):267-282. doi: 10.1007/s13238-018-0506-y. Epub 2018 Jan 17. PMID 29344809
- [Derived] Yan J, Zhang W, Feng Y, Liu X, Niu L, Guo Y, Zhou L, Shi M, Di C, Zhang Q, Wang X, Zhou J, Dai R, Ni L, Bao Z, Yan T, Hu Y, Wang P, Zhang T, Zhou M, Zuo W, Qu J. Autologous transplantation of P63+ lung progenitor cells in patients with bronchiectasis: A randomized, single-blind, controlled trial. Cell Rep Med. 2024 Nov 19;5(11):101819. doi: 10.1016/j.xcrm.2024.101819. PMID 39566467